CLINICAL TRIAL: NCT06835608
Title: Effects of Schroth-Based Three-Dimensional Exercise Program on Angle of Kyphosis, Muscle Strength, Balance, Pain, and Quality of Life in Patients With Postural Hyperkyphosis With Chronic Neck Pain
Brief Title: Effects of Schroth-Based Exercise on Kyphosis Angle, Muscle Strength, Balance, Pain, and Quality of Life in Hyperkyphosis With Chronic Neck Pain
Acronym: Kyphosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Collaborators: Baskent University Ankara Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA24/125
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Postural Kyphosis; Chronic Neck Pain
Keywords: postural hyperkyphosis; chronic neck pain

STUDY DESIGN:
Intervention Model Description: The study consists of two groups. Group 1 : exercise group Group 2: Control group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- three-dimensional schroth exercise group (Experimental): Schroth therapy, a three-dimensional exercise therapy program was developed in Germany in the 1920s by Katharina Schroth. The three-dimensional exercise program refers to the sagittal, frontal and horizontal planes. The three- dimensional Schroth exercise training consists of spinal lengthening and positional correction of the cervical, thoracic and lumbar regions in the sagittal plane, special breathing techniques and re-education of the neuromuscular system to improve kyphotic posture.
  Interventions: Other: Schroth Exercise Group
- corrective exercises for posture (Active Comparator): Corrective exercise program for posture will consist of deep neck flexor muscle strengthening exercises, lower and middle trapezius strengthening, neck isometric exercises.
  Interventions: Other: Postural Exercises Group

INTERVENTIONS:
Other: Schroth Exercise Group — The study group will receive electrotherapy treatment (hot pack, ultrasound, tens) to the neck area for 30 minutes in each session. After electrotherapy treatment, kyphotic posture correction exercises will be applied with the help of proprioceptive and extroceptive stimuli in the sagittal plane with mirror control and specific corrective breathing. In the exercise program, exercise practices will be performed in specific positions in supine, prone, sitting and standing. The exercise program will be planned for approximately 40 minutes in each session. A total of 20 sessions of electrotherapy and exercise will be performed for 4 weeks. At the end of the 4th week, after the electrotherapy sessions are completed, exercise applications will continue for the other 4 weeks by the physiotherapist who performs the exercise 3 days a week.
  Arms: three-dimensional schroth exercise group
Other: Postural Exercises Group — Patients to be included in the control group will receive electrotherapy treatment (ultrasound, tens, hotpack) to the neck area for 30 minutes in each session. After the electrotherapy treatment, posture corrective exercises will be applied. Corrective exercise program for posture will consist of deep neck flexor muscle strengthening exercises, lower and middle trapezius strengthening, neck isometric exercises. All strengthening exercises will be given 3 sets of 10 repetitions per day, each repetition for 10 seconds. Stretching exercises will be given to the shortened upper trapezius and pectoralis major muscles. Stretching exercises will be given 2 sets of 5 repetitions per day, with each repetition lasting 20 seconds. In the first 4 weeks, a total of 20 sessions of electrotherapy and exercise will be performed in corrective exercises for posture. At the end of the 4th week, exercise applications will continue for the other 4 weeks 3 days a week.
  Arms: corrective exercises for posture

SUMMARY:
The normal thoracic kyphosis angle of the spine is 20-40°, however, an angle of more than 40° is referred to as postural kyphosis, increased kyphosis or hyperkyphosis. Although postural kyphosis negatively affects individuals' general health status, physical performance, and quality of life, there is still no standardized protocol for correcting the thoracic kyphosis angle. Conservative treatment approaches such as postural training and exercises, manual therapy, postural corrective kinesiotaping, and orthotic use have been recommended for managing increased thoracic kyphosis. While numerous studies have demonstrated the effectiveness of three-dimensional exercise programs in the treatment of scoliosis, research examining their impact on kyphosis remains considerably limited.Nevertheless, the potential of these exercises to promote neuromuscular reorganization suggests that they may be similarly effective in individuals with thoracic kyphosis. This randomized controlled trial aims to evaluate the effects of a Schroth-based three-dimensional exercise program on kyphosis angle, trunk muscle strength, balance, pain, and quality of life in individuals with postural hyperkyphosis and chronic neck pain.

DETAILED DESCRIPTION:
Increasing thoracic kyphosis, spinal extensor muscle weakness, decreased spinal extension mobility, lumbo-pelvic pain, muscle activation and displacement of the scapula with changing traction angles have been associated with postural changes. It is evident that such alterations in posture have a biomechanical effect on the cervical and lumbar vertebrae. The presence of thoracic dysfunction has been documented in individuals experiencing chronic neck pain. Increases in both the thoracic kyphosis angle and flexor posture have been demonstrated to result in anterior displacement of the central gravity line. Displacement of the body's centre of gravity anteriorly has the potential to exert adverse effects on postural control.The association between postural changes and spinal extensor muscle weakness, increased kyphotic posture, decreased spinal extension mobility, lumbo-pelvic pain, muscle activation and displacement of the scapula with changing traction angles has been demonstrated. These postural changes have been demonstrated to exert a detrimental effect on postural stability, back pain, physical performance and quality of life.

The present study was meticulously designed as a Schroth-based three-dimensional exercise group and a control group, with a duration of eight weeks. The two groups will both undergo a programme comprising 20 sessions of electrotherapy and exercise, to be administered over a period of four weeks. Subsequent to the completion of the fourth week of electrotherapy sessions, the exercise applications will be continued for a further four weeks by the physiotherapist responsible for the study, who will undertake the programme three days per week. The intervention will consist of a series of educational sessions focusing on the development of postural perception, with a particular emphasis on the identification of postural kyphosis and the adoption of optimal posture in daily living. These educational sessions will be administered to both groups. The training programme will be delivered in a practical manner by the physiotherapist. A brochure will be provided to patients, serving as a reference guide for the exercises and considerations.

ELIGIBILITY:
Inclusion Criteria:

* Thoracic kyphosis angle > 45 degrees,
* Aged between 20 and 50 years,
* Have neck pain for more than 3 months,
* Neck pain visual analogue scale > 3,
* Not being treated for postural kyphosis in the last 6 months,
* Has no systemic disease

Exclusion Criteria:

* History of trauma or surgery on spinal joints,
* Participants with rheumatological and metabolic disorders,
* Participants with congenital postural deformity and scoliosis

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08-23 (Estimated)

PRIMARY OUTCOMES:
Angle of thoracic kyphosis | Baseline,4th week, 8th week
  The kyphosis angles of the participants will be measured using a flexible ruler and an inclinometer.As stated in the literature, thoracic kyphosis will be measured from C7-T12 spinal processes.Prior to molding the flexicurve ruler to the subject's spine, the C7 and T12 posterior spinous processes were located via palpation.The flexicurve ruler was then molded over the spine midline from C7 to T12. The resulting curve was traced on paper, and the locations of the C7 and T12 processes were labelled. The measurement was performed while the participant stood in a neutral upright posture with feet shoulder-width apart.The flexible ruler will be placed on the marked reference points. It will then be placed on the millimetrically divided paper without distorting its shape. The angular value of the curvature drawn on the paper from the contour of the flexible ruler will then be calculated. Another kyphosis angle will be measured by the same procedure using an inclinometer.

SECONDARY OUTCOMES:
Trunk Muscle Strength | Baseline,4th week, 8th week
  In our study, trunk extensor and flexor muscle strengths of participants will be measured with a hand-held dynamometer (Lafayette hand-held dynamometer model 01165 JTech, USA). Trunk extension strength will be measured in a prone position. The dynamometer will be positioned at the T4 level of the subjects, with the measurement being taken perpendicular to the body. Participants will be asked to assume the supine position with their knees straight, in order to measure the strength of their trunk flexor muscles. The dynamometer will be placed at the sternum level, and the measurement will be taken perpendicular to the trunk.Participants will be asked to cross their hands over their chest. In both measurements, participants are instructed to generate an isometric trunk extension force for a duration of two seconds, followed by a maximum isometric hold for five seconds. This measurement is then repeated on three occasions.
Balance Assessment | Baseline,4th week, 8th week
  Tetrax posturography device (Tetrax Potable Multiple System, Tetrax Ltd., Ramat Gan, Israel) is a device that allows objective assessment and recording of postural stability and fall risk.The measurements will be conducted in eight different positions: eyes open and closed with the head in a neutral position, eyes open and closed while standing on a foam surface with the head in a neutral position, eyes closed with the head rotated to the right and left, and eyes closed with the neck in full extension and flexion positions. The general stability index (SI) is to be conducted, with the displacement of each case's centre of mass and anterior-posterior weight distribution measurements being the basis on which it is to be assessed.
Spinal Stabilisation Activity | Baseline,4th week, 8th week
  The assessment of spinal stabilisation activity will be conducted utilising the Stabiliser Pressure Biofeedback device (PBU; Chattanooga Group-Australia).The pressure biofeedback device is a practical tool commonly used in clinical settings to measure the pressure generated during the activation of the Transversus Abdominis and Multifidus muscles, emphasizing segmental stabilization. The pressure gauge of the device ranges from 0 to 200 mmHg and is connected to an inflation unit (manometer). The measurement will be conducted with the patient in the prone position. The inflation unit of the device will be placed under the patient's umbilicus, positioned above the ASIS (anterior superior iliac spines). Before asking the patient to perform any muscle movement, the device's pressure will be set to 70 mmHg. Participants will be instructed to take a deep breath and gently draw the umbilicus toward the lumbar vertebrae, maintaining this position for 10 seconds
Visual Analogue Scale (VAS) | Baseline,4th week, 8th week
  The VAS (Visual Analogue Scale) will be utilised to evaluate the severity of neck pain. The patient will be requested to indicate the intensity of discomfort experienced over the preceding seven days on a 10-centimetre ruler that has been segmented into equal divisions. A score of 0 indicates an absence of pain, while a score of 10 represents the most severe pain. The measurement results will be used to assess the pain intensity.
Occiput Wall and Tragus Wall Distance | Baseline,4th week, 8th week
  To determine the anterior tilt of the head, the Tragus-to-Wall Distance will be measured. The participants should stand upright with their heels and back against the wall, maintaining a neutral neck position and closed chin. The distances between the occiput and the wall, as well as the tragus and the wall, will be measured using a tape measure in the sagittal plane. The average of these two measurements will then be calculated and recorded in centimetres.
Neck Disability Index | Baseline,4th week, 8th week
  The Neck Disability Index (NDI) is a self-reported questionnaire designed to assess neck pain-related disability. It consists of 10 items addressing daily activities such as personal care, lifting, reading, work, driving, sleeping, recreational activities, pain intensity, concentration, and headache. Each item is scored on a 6-point Likert scale ranging from 0 (no disability) to 5 (complete disability). The total score is calculated by summing the scores of all items and multiplying by two, resulting in a final score ranging from 0 to 100, where higher scores indicate a greater level of disability. In this study, the NDI will be used to evaluate neck-related functional limitations of participants, with scores expressed as a percentage of maximum possible disability.
Assessment of Quality of Life | Baseline,4th week, 8th week
  The Scoliosis Research Society-22 (SRS-22) Questionnaire is a widely accepted, simple, and practical tool developed by the Scoliosis Research Society to assess health-related quality of life in individuals with spinal deformities. In this study, the SRS-22 will be used to evaluate the quality of life of participants. The The questionnaire consists of 22 items grouped into five domains: pain, self-image/appearance, function/activity, mental health, and satisfaction with treatment. Each item is scored on a 5-point Likert scale, ranging from 1 (worst outcome) to 5 (best outcome). The total score is calculated by averaging the item scores within each domain or across all items. Higher scores reflect better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Tuğçe BAYRAM ERKOYUNCU, Study Chair — Baskent University; Hayri Baran YOSMAOĞLU, Prof., Study Director — Baskent University; Selin ÖZEN, Assoc. prof., Principal Investigator — Baskent University
Locations (1):
- Baskent University Umitkoy Outpatient Clinic, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data (IPD). However, once statistical analyses of all data are completed, aggregated results and summary statistical findings will be made available to researchers. These results will be shared in a de-identified format to ensure participant privacy. Interested researchers can request access to the results by contacting the principal investigator at (bayramtugce91@gmail.com)

REFERENCES:
- [Background] Bulut D, Dilek B, Kilinc A, Ellidokuz H, Oncel S. An investigation into the effects of kinesiotaping for posture correction on kyphosis angle, pain, and balance in patients with postmenopausal osteoporosis-associated thoracic kyphosis. Arch Osteoporos. 2019 Aug 13;14(1):89. doi: 10.1007/s11657-019-0634-x. PMID 31410649
- [Result] Alanay A, Cil A, Berk H, Acaroglu RE, Yazici M, Akcali O, Kosay C, Genc Y, Surat A. Reliability and validity of adapted Turkish Version of Scoliosis Research Society-22 (SRS-22) questionnaire. Spine (Phila Pa 1976). 2005 Nov 1;30(21):2464-8. doi: 10.1097/01.brs.0000184366.71761.84. PMID 16261127
- [Result] Telci EA, Karaduman A, Yakut Y, Aras B, Simsek IE, Yagli N. The cultural adaptation, reliability, and validity of neck disability index in patients with neck pain: a Turkish version study. Spine (Phila Pa 1976). 2009 Jul 15;34(16):1732-5. doi: 10.1097/BRS.0b013e3181ac9055. PMID 19770615
- [Result] Crasto CFB, Montes AM, Carvalho P, Carral JMC. Pressure biofeedback unit to assess and train lumbopelvic stability in supine individuals with chronic low back pain. J Phys Ther Sci. 2019 Oct;31(10):755-759. doi: 10.1589/jpts.31.755. Epub 2019 Oct 19. PMID 31645801
- [Result] Akkaya N, Doganlar N, Celik E, Aysse SE, Akkaya S, Gungor HR, Sahin F. TEST-RETEST RELIABILITY OF TETRAX(R) STATIC POSTUROGRAPHY SYSTEM IN YOUNG ADULTS WITH LOW PHYSICAL ACTIVITY LEVEL. Int J Sports Phys Ther. 2015 Nov;10(6):893-900. PMID 26618068
- [Result] De Blaiser C, De Ridder R, Willems T, Danneels L, Roosen P. Reliability and validity of trunk flexor and trunk extensor strength measurements using handheld dynamometry in a healthy athletic population. Phys Ther Sport. 2018 Nov;34:180-186. doi: 10.1016/j.ptsp.2018.10.005. Epub 2018 Oct 12. PMID 30366246
- [Result] Amatachaya P, Wongsa S, Sooknuan T, Thaweewannakij T, Laophosri M, Manimanakorn N, Amatachaya S. Validity and reliability of a thoracic kyphotic assessment tool measuring distance of the seventh cervical vertebra from the wall. Hong Kong Physiother J. 2016 Jul 13;35:30-36. doi: 10.1016/j.hkpj.2016.05.001. eCollection 2016 Dec. PMID 30931031
- [Result] Hunter DJ, Rivett DA, McKiernan S, Weerasekara I, Snodgrass SJ. Is the inclinometer a valid measure of thoracic kyphosis? A cross-sectional study. Braz J Phys Ther. 2018 Jul-Aug;22(4):310-317. doi: 10.1016/j.bjpt.2018.02.005. Epub 2018 Mar 6. PMID 29576490
- [Result] Greendale GA, Nili NS, Huang MH, Seeger L, Karlamangla AS. The reliability and validity of three non-radiological measures of thoracic kyphosis and their relations to the standing radiological Cobb angle. Osteoporos Int. 2011 Jun;22(6):1897-905. doi: 10.1007/s00198-010-1422-z. Epub 2010 Oct 12. PMID 20938766
- [Result] Barrett E, McCreesh K, Lewis J. Intrarater and interrater reliability of the flexicurve index, flexicurve angle, and manual inclinometer for the measurement of thoracic kyphosis. Rehabil Res Pract. 2013;2013:475870. doi: 10.1155/2013/475870. Epub 2013 Dec 12. PMID 24396603
- [Result] Lafage R, Steinberger J, Pesenti S, Assi A, Elysee JC, Iyer S, Lenke LG, Schwab FJ, Kim HJ, Lafage V. Understanding Thoracic Spine Morphology, Shape, and Proportionality. Spine (Phila Pa 1976). 2020 Feb 1;45(3):149-157. doi: 10.1097/BRS.0000000000003227. PMID 31513104
- [Result] Ozdemir Gorgu S, Algun ZC. A randomized controlled study of the effect of functional exercises on postural kyphosis: Schroth-based three-dimensional exercises versus postural corrective exercises. Disabil Rehabil. 2023 Jun;45(12):1992-2002. doi: 10.1080/09638288.2022.2083244. Epub 2022 Jun 12. PMID 35694970
- [Result] Bezalel T, Kalichman L. Improvement of clinical and radiographical presentation of Scheuermann disease after Schroth therapy treatment. J Bodyw Mov Ther. 2015 Apr;19(2):232-7. doi: 10.1016/j.jbmt.2014.04.008. Epub 2014 Apr 18. PMID 25892377
- [Result] Lehnert-Schroth C. Introduction to the Three-dimensional Scoliosis Treatment According to Schroth. Physiother (United Kingdom). 1992;78(11):810-815.
- [Result] Bansal S, Katzman WB, Giangregorio LM. Exercise for improving age-related hyperkyphotic posture: a systematic review. Arch Phys Med Rehabil. 2014 Jan;95(1):129-40. doi: 10.1016/j.apmr.2013.06.022. Epub 2013 Jul 9. PMID 23850611
- [Result] Bennell K, Khan K, McKay H. The role of physiotherapy in the prevention and treatment of osteoporosis. Man Ther. 2000 Nov;5(4):198-213. doi: 10.1054/math.2000.0369. PMID 11052899
- [Result] Kamali F, Shirazi SA, Ebrahimi S, Mirshamsi M, Ghanbari A. Comparison of manual therapy and exercise therapy for postural hyperkyphosis: A randomized clinical trial. Physiother Theory Pract. 2016;32(2):92-7. doi: 10.3109/09593985.2015.1110739. Epub 2016 Feb 10. PMID 26863146
- [Result] Perriman DM, Scarvell JM, Hughes AR, Lueck CJ, Dear KB, Smith PN. Thoracic hyperkyphosis: a survey of Australian physiotherapists. Physiother Res Int. 2012 Sep;17(3):167-78. doi: 10.1002/pri.529. Epub 2011 Dec 30. PMID 22223616
- [Result] Kado DM, Huang MH, Barrett-Connor E, Greendale GA. Hyperkyphotic posture and poor physical functional ability in older community-dwelling men and women: the Rancho Bernardo study. J Gerontol A Biol Sci Med Sci. 2005 May;60(5):633-7. doi: 10.1093/gerona/60.5.633. PMID 15972617
- [Result] Dolphens M, Cagnie B, Coorevits P, Vanderstraeten G, Cardon G, D'hooge R, Danneels L. Sagittal standing posture and its association with spinal pain: a school-based epidemiological study of 1196 Flemish adolescents before age at peak height velocity. Spine (Phila Pa 1976). 2012 Sep 1;37(19):1657-66. doi: 10.1097/BRS.0b013e3182408053. PMID 22108378
- [Result] Paine RM, Voight M. The role of the scapula. J Orthop Sports Phys Ther. 1993 Jul;18(1):386-91. doi: 10.2519/jospt.1993.18.1.386. PMID 8348140
- [Result] Fernandes VLS, Ribeiro DM, Fernandes LC, et al. de. Postural changes versus balance control and falls in community-living older adults: a systematic review. Fisioter em Mov. 2018; 31:25-31.
- [Result] Eum R, Leveille SG, Kiely DK, Kiel DP, Samelson EJ, Bean JF. Is kyphosis related to mobility, balance, and disability? Am J Phys Med Rehabil. 2013 Nov;92(11):980-9. doi: 10.1097/PHM.0b013e31829233ee. PMID 23636086
- [Result] Fernandes VLS, Ribeiro DM, Fernandes LC, Menezes RL de. Postural changes versus balance control and falls in community-living older adults: a systematic review. Fisioter em Mov. 2018;31(0):25-31
- [Result] Joshi S, Balthillaya G, Neelapala YVR. Thoracic Posture and Mobility in Mechanical Neck Pain Population: A Review of the Literature. Asian Spine J. 2019 Jun 3;13(5):849-860. doi: 10.31616/asj.2018.0302. Print 2019 Oct. PMID 31154701
- [Result] Jull GA, O'Leary SP, Falla DL. Clinical assessment of the deep cervical flexor muscles: the craniocervical flexion test. J Manipulative Physiol Ther. 2008 Sep;31(7):525-33. doi: 10.1016/j.jmpt.2008.08.003. PMID 18804003
- [Result] Lau KT, Cheung KY, Chan KB, Chan MH, Lo KY, Chiu TT. Relationships between sagittal postures of thoracic and cervical spine, presence of neck pain, neck pain severity and disability. Man Ther. 2010 Oct;15(5):457-62. doi: 10.1016/j.math.2010.03.009. PMID 20430685
- [Result] Oxland TR. Fundamental biomechanics of the spine--What we have learned in the past 25 years and future directions. J Biomech. 2016 Apr 11;49(6):817-832. doi: 10.1016/j.jbiomech.2015.10.035. Epub 2015 Nov 30. PMID 26706717
- [Result] Ludewig PM, Reynolds JF. The association of scapular kinematics and glenohumeral joint pathologies. J Orthop Sports Phys Ther. 2009 Feb;39(2):90-104. doi: 10.2519/jospt.2009.2808. PMID 19194022
- [Result] Katzman WB, Wanek L, Shepherd JA, Sellmeyer DE. Age-related hyperkyphosis: its causes, consequences, and management. J Orthop Sports Phys Ther. 2010 Jun;40(6):352-60. doi: 10.2519/jospt.2010.3099. PMID 20511692
- [Result] Young M, Michael L 2003 A review on postural realignment and its muscular and neural components. Elite Track, http://elitetrack.com
- [Result] Feng Q, Wang M, Zhang Y, Zhou Y. The effect of a corrective functional exercise program on postural thoracic kyphosis in teenagers: a randomized controlled trial. Clin Rehabil. 2018 Jan;32(1):48-56. doi: 10.1177/0269215517714591. Epub 2017 Jun 14. PMID 28610442
- [Result] Awad MA, Allah AH 2012 Relationship between thoracic kyphosis and trunk length in adolescence females. Journal of American Science 8: 580-583.
- [Result] Seidi F, Rajabi R, Ebrahimi I, Alizadeh MH, Minoonejad H. The efficiency of corrective exercise interventions on thoracic hyper-kyphosis angle. J Back Musculoskelet Rehabil. 2014;27(1):7-16. doi: 10.3233/BMR-130411. PMID 23948845
- [Result] Yang L, Lu X, Yan B, Huang Y. Prevalence of Incorrect Posture among Children and Adolescents: Finding from a Large Population-Based Study in China. iScience. 2020 May 22;23(5):101043. doi: 10.1016/j.isci.2020.101043. Epub 2020 Apr 8. PMID 32330860
- [Result] Vaughn DW, Brown EW 2007 The influence of an in-home based therapeutic exercise program on thoracic kyphosis angles. Journal of Back and Musculoskeletal Rehabilitation 20: 155-165.